CLINICAL TRIAL: NCT05677295
Title: Comparisons of the Impact of Duloxetine Versus Imipramine on Therapeutic Efficacy in Women With Stress Urinary Incontinence: a Randomized Controlled Study.
Brief Title: Therapeutic Efficacy in Women With Stress Urinary Incontinence
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Principal Investigator, Sheng-Mou Hsiao, Chief and Professor, Department of Obstetrics and Gynecology, Far Eastern Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 111220-F
Record Dates: First submitted 2023-01-01; First posted 2023-01-10 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2023-04

CONDITIONS: Women With Stress Urinary Incontinence
MeSH Terms: interventions — Duloxetine Hydrochloride; Imipramine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Duloxetine (Experimental)
  Interventions: Drug: duloxetine
- Imipramine (Active Comparator)
  Interventions: Drug: Imipramine

INTERVENTIONS:
Drug: duloxetine — Duloxetine 30 mg per day
  Arms: Duloxetine
Drug: Imipramine — Imipramine 25 mg per day
  Arms: Imipramine

SUMMARY:
We will get the impact of duloxetine versus imipramine on therapeutic efficacy in women with SUI.

DETAILED DESCRIPTION:
Background/Purpose: Pharmacologic treatments for female stress urinary incontinence (SUI) include duloxetine and imipramine. Duloxetine and Imipramine has been reported to have clinical significant therapeutic efficacy on female SUI and overactive bladder syndrome. However, there was no randomized controlled study to compare duloxetine and imipramine for the treatment of female SUI.

Patients and Methods: We will perform a prospective randomized controlled study to recruit 90 female SUI patients at the Obstetrics & Gynecology outpatient clinic of Far Eastern Memorial Hospital. All SUI female patients will be asked to complete ICIQ-UI, USS, OABSS, and bladder diary before and after 4 weeks' duloxetine versus imipramine treatment.

ELIGIBILITY:
Inclusion Criteria:

* Female patients over 25 years old with stress urinary incontinence.
* Patients who are currently not considered for surgical treatment.
* Patients who have undergone regular Kegel exercises but have poor results.

Exclusion Criteria:

* The result of urodynamic examination, if the main cause of urinary incontinence is detrusor overactivity.
* Those who are taking or plan to take monoamine oxidase inhibitor (MAOI) inhibitors.
* Patients with acute myocardial infarction.
* Those who are allergic to duloxetine, imipramine and dibenzazepine tricyclic antidepressants.
* Patients with uncontrolled narrow-angle glaucoma.
* Pregnant women.
* Those who are contraindicated to duloxetine or imipramine.
* Patients with suicidal ideation and behavior.

Min Age: 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-04-18 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Improvement of stress urinary incontinence | 4 weeks
  Urinary Incontinence Questionnaire (by ICIQ-UI short form)

SECONDARY OUTCOMES:
Improvement of urgency symptoms | 4 weeks
  Urgency severity scale
Improvement of overactive bladder symptoms | 4 weeks
  Overactive bladder symptom score

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Obstetrics and Gynecology, Far Eastern Memorial Hospital, Banqiao District, New Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No